CLINICAL TRIAL: NCT03671876
Title: Improving the Mobility of Patients After a Stroke (at a Sub-acute Stage) With the Help of the Selfit System - Testing the System's Feasibility, From the Point of View of the Therapist and the Patient.
Brief Title: Evaluation of Improvement in Mobility Skills for Sub-acute Stroke Patients, Using the Selfit System.
Acronym: Selfit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selfit Medical (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-08-ID-052717-CTIL; MOH_2018-04-11_002309 (Registry Identifier: Ministry of Health Israel)
Record Dates: First submitted 2018-09-06; First posted 2018-09-14 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: Stroke; Sub-acute; Mobility; Movement therapy; Exercise
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Methods; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention plus therapy (Active Comparator): Case group:
  A population that suffered a stroke and treated to improve mobility with the Selfit system (25 patients) for twice a week, at least 30 minutes per session, for a period of 3 weeks.
  Intervention with the Selfit system include a set of mobility task exercises.
  Interventions: Device: Intervention plus therapy
- Therapy and no intervention (No Intervention): Control group:
  A population that suffered a stroke and is being treated in the hospital without any interventions with the Selfit system.

INTERVENTIONS:
Device: Intervention plus therapy — Task oriented exercise plan to improve mobility for stroke patients
  Arms: Intervention plus therapy

SUMMARY:
Stroke is a leading cause of mobility disability for adults. Selfit is an advanced practice system that enables a wide range of exercises to improve patient mobility in the sub-acute stage after a stroke. The system collects, measures and analyzes the patient's activity in practice.

DETAILED DESCRIPTION:
Objectives of the study: An evaluation of the improvement of mobility after a stroke using the Selfit system.

Type of study: Case Control Study. Study population: 30 patients, after stroke (men and women aged 18-85). Criteria for Inclusion: Stroke patients who are capable to walk with a little help or no help at all, with or without any assitive device, for a distance of 10 meters.

Intervention: Random distribution of the study participants into two groups - Case: stroke patients (15 patients) - evaluation of patients using Selfit for 2 sessions per week, for a period of at least 30 minutes per session, during 3 weeks.

Control: Stroke patients (15 patients) - continuing with current therapy with no use of the Selfit system.

Measurement tools and outcome measures:

Duration of each treatment session, the duration of the actual treatment, the number of technical failures in the system during the exercise and the duration of each session will be recorded. At the end of the intervention, questionnaires describing the experience of using the system will be completed with a rating of the degree of satisfaction, convenience and simplicity of using the Selfit system. The following tests will be carried out : 10 meter walk test, Timed up and go test, Dynamic Gait Index (DGI).

Analysis of the data: For each patient's treatment, a personal activity profile will be established that includes the timing and speed of walking, the number of steps, the length and width of each step, the elevation of the leg at each step and the accuracy of the patient's performance. Statistical analysis will examine the various levels of activity throughout the intervention period for each patient and for the entire study population before and after the intervention. At the same time, the correlation between the level of activity in the treatment and the scores on the neurological tests will be examined. The data will be presented descriptively for the therapist and patient. For statistical analysis, the SPPS version 21 (IBM) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Stroke .Must walk with little or no help at all, with or without an assistive device, for a distance of at least 10 meters.

Exclusion Criteria:

- .Patients suffering from significant lower back pain and / or previous orthopedic impairment and / or cognitive impairment (grade 18 and below according to the MOCA test).

.Patients who are unable to move with little or no help at all, with or without an assistive device, for a distance of 10 meters.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in patient's average speed | 3 weeks
  Change from baseline in mobility skills - speed (m/sec)
Changes in patient's average distance | 3 weeks
  Change from baseline in mobility skills - distance (m)
Changes in patient's number of steps | 3 weeks
  Change from baseline in mobility skills - number of steps
Changes in patient's steps height | 3 weeks
  Change from baseline in mobility skills - steps height (avg. in cm)

CONTACTS AND LOCATIONS:
Overall Officials: Israel Dudkiewicz, Prof., Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel